CLINICAL TRIAL: NCT00040989
Title: Phase II Study of BAY 56-3722 in Patients With Recurrent, Unresectable, or Metastatic Renal Cell Carcinoma
Brief Title: BAY 56-3722 in Treating Patients With Recurrent, Unresectable, or Metastatic Kidney Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: UCLA-0201019; CDR0000069432 (Registry Identifier: PDQ (Physician Data Query)); UTHSC-0125011152; BAYER-100364; NCI-G02-2090
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2006-12

CONDITIONS: Stage IV Renal Cell Cancer; Recurrent Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — 20-O-(Nalpha-(4-(3-O-methylfucopyranosyloxy)phenylaminothiocarbonyl)histidylvalyl)camptothecin

INTERVENTIONS:
Drug: BAY 56-3722
Procedure: enzyme inhibitor therapy

SUMMARY:
RATIONALE: BAY 56-3722 may stop the growth of cancer cells by blocking the enzymes necessary for tumor cell growth.

PURPOSE: Phase II trial to study the effectiveness of BAY 56-3722 in treating patients who have recurrent, unresectable, or metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the tumor response rate of patients with recurrent, unresectable, or metastatic renal cell carcinoma treated with BAY 56-3722.
* Determine the duration of response, time to progression, and survival of patients treated with this drug.
* Determine the qualitative and quantitative toxic effects of this drug in these patients.
* Determine the pharmacokinetics of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive BAY 56-3722 IV over 30 minutes on days 1-3. Treatment repeats every 3 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 6 months.

PROJECTED ACCRUAL: A total of 20-140 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed renal cell carcinoma (RCC)
* Recurrent AND unresectable disease OR
* Unresectable disease OR
* Metastatic disease
* At least 1 bidimensionally measurable lesion by CT scan or MRI
* No metastatic brain or meningeal tumors unless more than 3 months since prior surgery and/or gamma knife radiosurgery, 2 subsequent negative imaging studies at least 4 weeks apart, clinically stable, and no concurrent corticosteroids or anticonvulsants

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9 g/dL

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST and ALT less than 2.5 times ULN (5 times ULN if liver metastases present)
* No chronic hepatitis B or C

Renal:

* Creatinine no greater than 1.5 mg/dL
* Calcium normal

Cardiovascular:

* No clinically evident congestive heart failure
* No serious cardiac arrhythmias
* No symptoms of coronary heart disease
* No symptoms of ischemia

Other:

* HIV negative
* No active infections requiring systemic antibacterial, antifungal, or antiviral therapy
* No other malignancy within the past 3 years except carcinoma in situ of the cervix, adequately treated basal cell carcinoma, or superficial bladder tumors (Ta, Tis, or T1)
* No substance abuse
* No medical, psychological, or social conditions that would preclude study
* No known or suspected allergy to study drug or any other study agents
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 6 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior anticancer vaccine therapy
* No prior bone marrow transplantation or stem cell rescue
* More than 4 weeks since prior thalidomide and bevacizumab
* At least 4 weeks since prior interleukin-2 and interferon
* No more than 2 prior regimens
* No concurrent bone marrow transplantation or stem cell rescue

Chemotherapy:

* No prior cytotoxic chemotherapy
* No concurrent cytotoxic chemotherapy

Endocrine therapy:

* See Disease Characteristics
* No prior hormonal therapy for RCC
* No concurrent hormonal therapy for RCC

Radiotherapy:

* See Disease Characteristics
* More than 4 weeks since prior radiotherapy
* No prior radiotherapy to indicator lesion unless progression is documented

Surgery:

* See Disease Characteristics
* More than 3 weeks since prior major surgery

Other:

* At least 4 weeks since prior investigational anticancer drugs
* No other concurrent investigational anticancer drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J. Gitlitz, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (26):
- United States (26):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Oncology-Hematology Group of South Florida, Miami, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of Rochester Medical Center, Rochester, New York
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Oregon Cancer Institute, Portland, Oregon
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas